CLINICAL TRIAL: NCT05594212
Title: The Effect of Abdominal Breathing on Improving of Depression, Anxiety, and Heart Rate Variability in Obstructive Sleep Apnea Patients With Depressive Symptoms
Brief Title: Abdominal Breathing for Depression, Anxiety, Heart Rate Variability in Obstructive Sleep Apnea Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Taipei University of Nursing and Health Sciences (Other)
Collaborators: Cheng-Hsin General Hospital (Other)
Responsible Party: Principal Investigator, Xuan-Yi Huang, RN, DNSc, Professor, National Taipei University of Nursing and Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: (879)110A-25
Record Dates: First submitted 2022-10-21; First posted 2022-10-26 (Actual); Last update posted 2022-10-26 (Actual); Status verified 2022-10

CONDITIONS: Obstructive Sleep Apnea
Keywords: abdominal breathing; obstructive sleep apnea; depression; anxiety; heart rate variability
MeSH Terms: conditions — Sleep Apnea, Obstructive; Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: This study method adopts an experimental research design and divided into experimental group and control group by random sampling. Experimental group receives abdominal breathing training, whereas control group without receiving abdominal breathing training.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The effectiveness of receiving abdominal breathing training (Experimental): The effectiveness of receiving abdominal breathing training Training for 8 weeks (1 time a week, 15 minutes each time). Performed one-on-one by a trainer in a sleep center. At home, you can use the abdominal breathing training video to train yourself (10 minutes a day, can be divided into 10 minutes), and you need to fill in the abdominal breathing training log.
  Interventions: Behavioral: Abdominal breathing training
- The effectiveness of not receiving abdominal breathing training (No Intervention): The effectiveness of not receiving abdominal breathing training The trainer does not provide abdominal breathing training, does not perform abdominal breathing exercises at home, and does not need to fill in abdominal breathing training logs.

INTERVENTIONS:
Behavioral: Abdominal breathing training — In the sleep center, it is carried out in a one-on-one manner by the trainer. At home, self-training through abdominal breathing training videos (10 minutes per day, you can accumulate up to 10 minutes in divided doses)
  Arms: The effectiveness of receiving abdominal breathing training

SUMMARY:
The research topic is to explore the effectiveness of abdominal breathing on improving of depression, anxiety, and heart rate variability in obstructive sleep apnea patients with depressive symptoms. This study method adopts an experimental research design and divided into experimental group and control group by random sampling. Experimental group receives abdominal breathing training, whereas control group without receiving abdominal breathing training.

DETAILED DESCRIPTION:
Obstructive Sleep Apnea (OSA) is a common chronic disease with frequent comorbidity of depression. When we use sedatives, antidepressants or hypnotics for the treatment of depression, these drugs may worsen symptoms of OSA leading to aggravation of original depressed moods. Therefore, the research topic is to explore the effectiveness of abdominal breathing on improving of depression, anxiety, and heart rate variability among obstructive sleep apnea patients with depressive symptoms. This study method adopts an experimental research design and divided into experimental group and control group by random sampling. Experimental group receives abdominal breathing training, whereas control group without receiving abdominal breathing training. The research is conducted with experimental and control groups. The effectiveness assessment will use the Beck Depression Inventory (BDI) Beck Anxiety Inventory (BAI) and check the heart rate variability (HRV). Both groups received the pre-test before the abdominal breathing training. The post-test was carried out at the fourth and eighth weeks of training. The experimental group is given abdominal breathing training for a total of 8 weeks, with the training in the hospital once a week, 15 minutes for each time, in combination with self-training at home under videos guidance for 10 minutes per day (10 minutes, for one time or several times accumulated) .The expected result is through abdominal breathing, the depression, anxiety, and heart rate variability of OSA patients with depressive symptoms can improve, and even with less use of medication.

ELIGIBILITY:
Inclusion Criteria:

* aged 20-64 years old.
* Be able to communicate with Chinese and Taiwanese, and who can express themselves without barriers.
* A person who is clearly conscious and can perform breathing exercises autonomously.
* Patients diagnosed with obstructive sleep apnea (AHI≧5) according to polysomnography and depression score ≧14 points measured by Beck Depression Inventory-II (Chinese version).

Exclusion Criteria:

* Patients with COPD.
* Patients with suicidal ideation.
* Obstructive sleep apnea AHI≧60.
* Those who have learned abdominal breathing.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2022-08-05 (Actual); Study Completion 2022-09-24 (Actual)

PRIMARY OUTCOMES:
Beck Depression Inventory-II | Pre-test
  The total items of Beck Depression Inventory-II are 21. The score of each item is from 0-3. The score 0-13 is the normal range, 14-19 is the mild depression, 20-28 is the moderate depression, and 29-63 is the severe depression.
Beck Depression Inventory-II | Post-test at week 4
  The total items of Beck Depression Inventory-II are 21. The score of each item is from 0-3. The score 0-13 is the normal range, 14-19 is the mild depression, 20-28 is the moderate depression, and 29-63 is the severe depression.
Beck Depression Inventory-II | Post-test at week 8
  The total items of Beck Depression Inventory-II are 21. The score of each item is from 0-3. The score 0-13 is the normal range, 14-19 is the mild depression, 20-28 is the moderate depression, and 29-63 is the severe depression.

SECONDARY OUTCOMES:
Beck anxiety inventory | Pre-test
  The total items of Beck anxiety inventory are 21. The score of each item is from 0-3. The score 0-7 is the least mild anxiety, 8-15 is the mild anxiety, 16-25 is the moderate anxiety, and 26-63 is the severe anxiety.
Beck anxiety inventory | Post-test at week 4
  The total items of Beck anxiety inventory are 21. The score of each item is from 0-3. The score 0-7 is the least mild anxiety, 8-15 is the mild anxiety, 16-25 is the moderate anxiety, and 26-63 is the severe anxiety.
Beck anxiety inventory | Post-test at week 8
  The total items of Beck anxiety inventory are 21. The score of each item is from 0-3. The score 0-7 is the least mild anxiety, 8-15 is the mild anxiety, 16-25 is the moderate anxiety, and 26-63 is the severe anxiety

OTHER OUTCOMES:
Heart rate variability | Pre-test
  Changes in heart rate variability measured by TS-0411
Heart rate variability | Post-test at week 4
  Changes in heart rate variability measured by TS-0411
Heart rate variability | Post-test at week 8
  Changes in heart rate variability measured by TS-0411

CONTACTS AND LOCATIONS:
Overall Officials: Xuan-Yi Huang, DNSc, Principal Investigator — National Taipei University of Nursing and Health Sciences
Locations (1):
- Xuan-Yi Huang, Taipei, Peitou, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Akberzie W, Hesselbacher S, Aiyer I, Surani S, Surani ZS. The Prevalence of Anxiety and Depression Symptoms in Obstructive Sleep Apnea. Cureus. 2020 Oct 27;12(10):e11203. doi: 10.7759/cureus.11203. PMID 33269134
- [Background] Asghari A, Mohammadi F, Kamrava SK, Tavakoli S, Farhadi M. Severity of depression and anxiety in obstructive sleep apnea syndrome. Eur Arch Otorhinolaryngol. 2012 Dec;269(12):2549-53. doi: 10.1007/s00405-012-1942-6. PMID 22298252
- [Background] Bollig SM. Encouraging CPAP adherence: it is everyone's job. Respir Care. 2010 Sep;55(9):1230-9. PMID 20800003
- [Background] Bordoni B, Purgol S, Bizzarri A, Modica M, Morabito B. The Influence of Breathing on the Central Nervous System. Cureus. 2018 Jun 1;10(6):e2724. doi: 10.7759/cureus.2724. PMID 30083485
- [Background] Chen YF, Huang XY, Chien CH, Cheng JF. The Effectiveness of Diaphragmatic Breathing Relaxation Training for Reducing Anxiety. Perspect Psychiatr Care. 2017 Oct;53(4):329-336. doi: 10.1111/ppc.12184. Epub 2016 Aug 23. PMID 27553981
- [Background] Senaratna CV, Perret JL, Lodge CJ, Lowe AJ, Campbell BE, Matheson MC, Hamilton GS, Dharmage SC. Prevalence of obstructive sleep apnea in the general population: A systematic review. Sleep Med Rev. 2017 Aug;34:70-81. doi: 10.1016/j.smrv.2016.07.002. Epub 2016 Jul 18. PMID 27568340
- [Background] Tsai SH, Wang MY, Miao NF, Chian PC, Chen TH, Tsai PS. CE: original research: The efficacy of a nurse-led breathing training program in reducing depressive symptoms in patients on hemodialysis: a randomized controlled trial. Am J Nurs. 2015 Apr;115(4):24-32; quiz 33, 42. doi: 10.1097/01.NAJ.0000463023.48226.16. PMID 25793429
- [Background] Zaccaro A, Piarulli A, Laurino M, Garbella E, Menicucci D, Neri B, Gemignani A. How Breath-Control Can Change Your Life: A Systematic Review on Psycho-Physiological Correlates of Slow Breathing. Front Hum Neurosci. 2018 Sep 7;12:353. doi: 10.3389/fnhum.2018.00353. eCollection 2018. PMID 30245619